CLINICAL TRIAL: NCT03732209
Title: A Remotely Delivered Episodic Future Thinking Intervention to Improve Management of Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Carilion Clinic (Other); University at Buffalo (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jeffrey Stein, Research Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2696; 1R21NR018349-01 (NIH)
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will engage in episodic future or control thinking in the natural environment. All participants will also receive case management regarding the Traffic Light Diet, modified for type 2 diabetes to include glycemic index of foods, as well as the Traffic Light Activity Plan and other techniques to aid in weight loss (e.g., self-monitoring).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants assigned to both groups will be masked to experimental hypotheses. Research personnel who will be conducting assessment sessions, including weight measurements, will not be informed of participants' group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic future thinking (Experimental): Participants will generate positive future events and related text cues that will be accessed via an electronic app to engage in episodic future thinking.
  Interventions: Behavioral: Episodic future thinking
- Control thinking (Sham Comparator): Participants will generate non-future-oriented information and related text cues that will be accessed via an electronic app to engage in control thinking..
  Interventions: Behavioral: Control Thinking

INTERVENTIONS:
Behavioral: Episodic future thinking — Participants will engage in episodic future thinking, prompted via text-based cues, when making decisions about dietary, exercise, and medication adherence choices.
  Arms: Episodic future thinking
Behavioral: Control Thinking — Participants will engage in non-future-oriented control thinking, prompted via text-based cues, when making decisions about dietary, exercise, and medication adherence choices.
  Arms: Control thinking

SUMMARY:
The goals of this project are to assess the efficacy of remotely delivered episodic future thinking for reducing delay discounting and improving management of type 2 diabetes, including glycemic control, weight loss, medication adherence, dietary intake, physical activity, and blood pressure. This will be accomplished by randomly assigning participants (N = 64) to episodic future thinking or control thinking groups, while tracking outcome measures before, during, and after the 4-month intervention, as well at a 6-month follow-up visit. Participants in both groups will also receive access to an information-based weight loss intervention.

DETAILED DESCRIPTION:
Participants (N = 64) will be randomly assigned to either an episodic future thinking group or control thinking groups. Participants will generate episodic future events or control information, as well as related text-based cues, and will be prompted via smartphone or web application to engage in episodic future or control thinking frequently in their natural environment (e.g., at home or work, before meal times, and in high-risk situations) for a 4-month period. Participants in both groups will be provided with one-on-one, phone-based case management and provided with instructional materials and behavioral tools for weight loss and diabetes management. Instructional materials will include: 1) a modified version of the Traffic Light Diet, which utilizes red, yellow, and green labels for food to guide participants toward the goal of consuming low energy dense, low glycemic, high nutrient dense foods; 2) the Traffic Light Activity Program, which also utilizes red, yellow, and green labels for different levels of caloric expenditure, and 3) tools for self-monitoring of weight, diet, and/or physical activity.

Participants will complete four laboratory-based assessment sessions in which the investigators assess body weight, height, waist and hip circumference, glycemic control (HbA1C), adherence to oral glucose-lowering medication, delay discounting, reinforcing efficacy of food, and blood pressure. These assessments will be completed before the intervention (Week 0), during the intervention (8 weeks), and immediately after the intervention (Week 16), as well after a 2-month post-intervention follow-up (Week 24). The latter three assessments sessions will also include questions to measure participants' perceived effectiveness and ease of use of the intervention. Participants will also complete several remote assessments, including dietary intake and physical activity (during Weeks 0, 8, and 16; via accelerometer), as well as delay discounting and reinforcing efficacy of food (during Weeks 3, 8, and 16).

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI of 25 or greater)
* Poorly controlled type 2 diabetes (HbA1C of 8% or greater)
* Prescribed or recommended oral glucose-lowering medication

Exclusion Criteria:

* Current insulin therapy for type 2 diabetes
* History of gestational diabetes
* Pregnant or lactating
* Not ambulatory
* Intellectual impairment
* Unmanaged medical or psychiatric disorder
* Abnormal glucose related to medications (e.g, glucocorticoids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Stein, PhD, Principal Investigator — Virginia Tech Carilion School of Medicine and Research Institute; John W Epling, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in person at the Fralin Biomedical Research Institute at Virginia Tech Carilion, from March 2019 to March 2020.
Pre-assignment Details: Participants were randomized to episodic future thinking and control groups at Week 3 of the study.
Period: Overall Study
Arm/Group | Episodic Future Thinking | Control Thinking
Started | 20 | 23
Completed | 8 | 10
Not Completed | 12 | 13
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Episodic Future Thinking | Control Thinking | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.38 (10.9) | 56.9 (13.1) | 54.89 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (kg/m^2)
  kg/m^2 | 38.46 (8.1) | 39.60 (6.5) | 38.96 (7.2)
hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — Hemoglobin A1c, a measure of glycemic control
  percentage of glycosylated hemoglobin | 9.58 (1.2) | 9.37 (2.3) | 9.48 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin
Description: Glycemic control will be assessed by change in glycosylated hemoglobin (hemoglobin A1C, or HbA1c), a standardized diagnostic measure for type 2 diabetes.
  Negative change scores indicate a reduction in percentage of glycosylated hemoglobin (improved glycemic control); positive scores indicate an increase in percentage of glycosylated hemoglobin (worsened glycemic control)
Time Frame: Baseline, 8 weeks, 16 weeks, and 24 weeks
Population: Participants randomized to groups at Week 3 of the study
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Episodic Future Thinking | Control Thinking
Number analyzed (Participants) | 8 | 10
percentage of glycosylated hemoglobin
  Week 8 | -1.2 (0.77) | -0.30 (0.63)
  Week 16: number analyzed (Participants) | 6 | 4
  Week 16 | -1.4 (1.59) | -0.5 (0.4)
  Week 24: number analyzed (Participants) | 4 | 4
  Week 24 | -3.3 (1.2) | -1 (1)
Statistical Analysis 1: Comparison: Episodic Future Thinking vs Control Thinking; Due to minimal data being available at Weeks 16 and 24 due to COVID-19-related attrition, only baseline (Week 0) and Week 8 data were included in the analysis; Test type: Superiority; p = .017, ANOVA — This p value reflects the interaction between group (episodic future thinking, control) and time (baseline, Week 8); F value, group x time interaction = 7.155 — Reported values in outcome measures data table reflect mean change in glycosylated hemoglobin for each group (Session 2 - Session 1)

2. Primary Outcome: Change in kg/m^2 (Body Mass Index)
Description: Change in kg/m^2 (body mass index) will be measures using a digital scale
  Negative scores indicate reductions in kg/m^2; positive scores indicate increases in BMI.
Time Frame: Baseline, 8 weeks, 16 weeks, and 24 weeks
Population: Participants randomized to groups at Week 3 of the study
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Episodic Future Thinking | Control Thinking
Number analyzed (Participants) | 8 | 10
kg/m^2
  Week 8 | -1.2 (0.81) | -0.3 (1.04)
  Week 16: number analyzed (Participants) | 6 | 4
  Week 16 | -1.4 (1.11) | 0.71 (0.61)
  Week 24: number analyzed (Participants) | 4 | 4
  Week 24 | -0.7 (0.96) | 0.1 (1.67)
Statistical Analysis 1: Comparison: Episodic Future Thinking vs Control Thinking; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .042, ANOVA — This p value reflects the interaction between group (episodic future thinking, control) and time (baseline, Week 8); F value, group x time interaction = 4.885 — The values reported in the outcome measures data table reflect mean change in AUC (Session 2 - Session 1)

3. Primary Outcome: Change in Delay Discounting Area Under the Curve (Normalized)
Description: Delay discounting will be assessed using a computerized task that assess participants' indifference points, or the objective amount of a smaller, immediate reward that is subjectively equivalent to a delayed, larger reward ($100), across a range of delays (1 month, 3 months, 6 months, 1 year, 3 years, 5 years, and 12 years). Indifference points will be expressed as a proportion of the larger reward (0 to 1). This delay discounting curve (indifference points as a function of delay) will be summarized using area under the curve (AUC), calculated using subjective value of the delayed reward (0 to 1) as the y-axis unit and delay as the x-axis unit. Individual delays are converted to ordinal units (1-7) prior to analysis. AUC is expressed as a proportion of the maximum possible AUC. This normalized measure of AUC varies from 0 (maximum discounting) to 1 (minimum discounting).
  Positive scores indicate reductions in delay discounting (i.e., increases in AUC across time); negative sco
Time Frame: Baseline, 8 weeks, 16 weeks, and 24 weeks
Population: Participants randomized to groups at Week 3
Measure: Mean (Standard Deviation); unit: Proportion of reward*ordinal delay
Arm/Group | Episodic Future Thinking | Control Thinking
Number analyzed (Participants) | 8 | 10
Proportion of reward*ordinal delay
  Week 8 | 0.07 (0.13) | -0.04 (0.12)
  Week 16: number analyzed (Participants) | 6 | 4
  Week 16 | 0.07 (0.18) | 0.02 (0.13)
  Week 24: number analyzed (Participants) | 4 | 4
  Week 24 | 0.15 (0.15) | -0.07 (0.24)
Statistical Analysis 1: Comparison: Episodic Future Thinking vs Control Thinking; Due to minimal data available at Week 16 and 24 due to COVID-19-related attrition, only ratings from Week 8 were included in the analysis; Test type: Superiority; p = .146, ANOVA — This p value reflects the interaction between group (episodic future thinking, control) and time (baseline, Week 8); F value, group x time interaction = 2.33

4. Secondary Outcome: Perceived Treatment Effectiveness
Description: Perceived treatment effectiveness for the EFT and control conditions will be measured using a 5-point scale, ranging from 1 (not at all) to 5 (extremely).
  Higher scores reflect greater perceived effectiveness.
Time Frame: 8 weeks, 16 weeks, and 24 weeks
Population: Participants randomized to groups at Week 3 of the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale of 1-5
Arm/Group | Episodic Future Thinking | Control Thinking
Number analyzed (Participants) | 8 | 10
score on a scale of 1-5
  Week 8 | 3.63 [3 to 4.25] | 2.4 [1.25 to 3]
  Week 16: number analyzed (Participants) | 6 | 4
  Week 16 | 3.5 [3 to 3.75] | 3 [2.5 to 4]
  Week 24: number analyzed (Participants) | 4 | 4
  Week 24 | 3 [3 to 3] | 3.75 [3.25 to 5]
Statistical Analysis 1: Comparison: Episodic Future Thinking vs Control Thinking; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .042, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.23

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 24-week participation period.
Arm/Group | Episodic Future Thinking | Control Thinking
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic caused a spike in attrition, with many of the n=59 participants who enrolled in the trial to not reach trial randomization in Week 3 and study completion in Week 24. Likewise, the long-lasting restrictions on in-person assessments and the lack of reliable and feasible methods to collect these measures remotely limited new enrollments. As a result, this trial did not meet its recruitment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03732209/Prot_SAP_000.pdf